CLINICAL TRIAL: NCT07029139
Title: A Multicenter, Randomized, Controlled, Open-label Phase II Clinical Study Evaluating the Efficacy and Safety of JMT601 Injection in Participants With Primary Membranous Nephropathy
Brief Title: A Study to Learn More About the Effects and Safety of JMT601 in Adults With Primary Membranous Nephropathy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JMT601-003
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Primary Membranous Nephropathy
MeSH Terms: interventions — Rituximab; Cyclosporine

STUDY DESIGN:
Intervention Model Description: This is a multi-center, randomized, controlled, open-label Phase II clinical study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- JMT601 (Part 1) (Experimental): JMT601
  Interventions: Drug: JMT601 Injection
- Rituximab (Part 1) (Active Comparator): Rituximab
  Interventions: Drug: JMT601 Injection; Drug: Cyclosporin Capsules
- JMT601 (Part 2) (Experimental): JMT601
  Interventions: Drug: Rituximab; Drug: Cyclosporin Capsules
- Cyclosporin Capsules (part 2) (Active Comparator): Cyclosporin Capsules
  Interventions: Drug: JMT601 Injection; Drug: Rituximab

INTERVENTIONS:
Drug: JMT601 Injection — In accordance with the protocol
  Arms: Cyclosporin Capsules (part 2); JMT601 (Part 1); Rituximab (Part 1)
Drug: Rituximab — In accordance with the protocol
  Arms: Cyclosporin Capsules (part 2); JMT601 (Part 2)
Drug: Cyclosporin Capsules — In accordance with the protocol
  Arms: JMT601 (Part 2); Rituximab (Part 1)

SUMMARY:
This study is a multicenter, randomized, controlled, open-label, Phase Ⅱ clinical study to evaluate the efficacy, safety, Pharmacokinetics characteristics, Pharmacodynamics effects, and immunogenicity of JMT601 in participants with primary membranous nephropathy.

The study has two parts. Part one is dose escalation part, and Part two is dose expansion part.

ELIGIBILITY:
Inclusion Criteria:

1. The age range is between 18 and 80 years old, regardless of gender.
2. Diagnosed with primary membranous nephropathy by renal biopsy during the screening/induction period or within 24 months before screening. Pathological reports must be reviewed by the investigator prior to study drug administration.
3. The glomerular filtration rate (eGFR) estimated by CKD-EPI formula is ≥ 40ml/min/1.73m^2, or the endogenous creatinine clearance rate (CrCl) based on 24-hour urine examination is ≥ 40ml/min.
4. Participants taking angiotensin converting enzyme inhibitors/angiotensin II receptor antagonists must maintain a stable dose for at least 4 weeks before screening;
5. Participants with systolic blood pressure ≤140 mmHg and diastolic blood pressure ≤ 90 mmHg at screening.
6. During the screening period and the baseline visit, the 24-hour urine protein is > 3.5g.
7. Have never received immunosuppressive therapy for PMN (cyclophosphamide, calcineurin inhibitors, such as cyclosporine and tacrolimus) and B cell exhaustion therapy (such as rituximab); or relapsed after receiving the above treatment to achieve complete remission or partial remission (comprehensively judged and recorded by the researcher), and have not received the above treatment after recurrence (excluding those who are ineffective or resistant to B cell depletion drugs).
8. Have fully understood this study and voluntarily signed the informed consent form.

Exclusion Criteria:

1. Secondary membranous nephropathy.
2. Diagnostic renal biopsy shows evidence of glomerular crescent formation, which suggests the diagnosis of other renal diseases or renal biopsy evidence of interstitial fibrosis/tubular atrophy in cortical area > 50%.
3. Uncontrolled blood pressure as judged by the investigator within the 3 months prior to screening.
4. Individuals with evidence of a ≥50% decrease in urine protein within the first 6 months before screening.
5. Currently undergoing or planning to undergo renal replacement therapy during the study period.
6. Type 1 diabetes or type 2 diabetes with diabetic nephropathy (confirmed by renal biopsy report) or without biopsy-confirmed diabetic nephropathy but with a diabetes duration ≥5 years.
7. Presence of severe, progressive, or uncontrolled comorbidities.
8. Individuals who have had or currently have malignant tumors.
9. Participants with autoimmune diseases requiring systemic immunosuppression therapy, or those judged by researchers to have autoimmune diseases that interfere with the clinical evaluation of primary membranous nephropathy or are not suitable for clinical trials.
10. A history of previous or current hemolytic anemia, Evans syndrome, arteritis.
11. Participants with suspected active or latent tuberculosis patients based on medical history or tuberculosis screening.
12. Severe active bacterial, viral, fungal, mycobacterial, parasitic, or other infections requiring systemic antibiotics or antiviral treatment within 1 month before screening.
13. Have received prescribed treatment for membranous nephropathy before screening.
14. Participants using of complementary therapies that may interfere with the investigator's assessment of participant efficacy and safety within 4 weeks prior to randomization.
15. Live vaccines or major surgery within 28 days before the investigational drug administration or undergoing major surgery.
16. Participants who have participated in clinical trials of other drugs with a screening time less than 30 days from the last administration or the five half-lives of the original drug (whichever is longer), or those who plan to participate in clinical trials of another drug during the study period.
17. Participants who have received targeted CD47 or signal regulatory protein α (SIRPα) therapy.
18. A history of alcoholism or drug abuse within 12 months.
19. Virology test results at screening meet the criteria:

    HBsAg positivity; If HBsAg is negative and HBcAb is positive, HBV DNA should be exceeding the upper limit of the local laboratory reference range; Positive hepatitis C virus (HCV) antibody with detectable HCV RNA; Positive serology for human immunodeficiency virus (HIV).
20. Any of the following abnormal laboratory test results during screening: hemoglobin<80g/L, platelet count<100× 10^9/L , absolute neutrophil count<1.5× 10^9/L , AST or ALT values>2× upper limit of normal (ULN), CD4+ T lymphocyte count < 300 cells/μL, QTcF>450 ms for males and >460 ms for females.
21. Participants who have previously shown resistance to CD20 inhibitors or cyclosporine.
22. Known history of severe hypersensitivity reactions to humanized monoclonal antibodies or documented allergy to any component of rituximab (dose-escalation part only), JMT601 injection, or cyclosporine (dose-expansion part only).
23. Pregnant or lactating women; Women of childbearing potential not undergoing sterilization who are unwilling to use adequate contraception during treatment and for at least 6 months after the last dose of the investigational drug.
24. Men not undergoing sterilization who are unwilling to use barrier contraception during the study and for at least 6 months after the last dose of the investigational drug, and who refuse to ensure their partners use additional contraceptive methods (e.g., oral contraceptives, intrauterine devices, barrier methods, or spermicides).
25. Other conditions that the investigator deems render the subject unsuitable for study participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events in Part 1 | Up to 24 weeks
Overall Remission Rate at week 52 in Part 2 | week 52
  Participants with overall remission are those achieving either complete remission or partial remission

SECONDARY OUTCOMES:
Blood drug concentration of JMT-601 in Part 1 | week 24
Immunological remission in the anti-PLA2R antibody positive population in Part 1 | week 12, 24
  Proportion of anti-PLA2R antibody-positive participants achieving immunological remission
Changes in anti-PLA2R antibody titers from baseline in anti-PLA2R antibody positive population in Part 1 | week 24
Overall Remission Rate in Part 1 | weeks 12, 24
Complete Remission Rate in Part 1 | weeks 12, 24
  A complete remission is defined as UPCR (based on 24-hour urine collection) ≤ 0.3, and a stable eGFR (remaining unchanged or decreasing by ≤ 15% compared with the baseline)
ADA (anti-drug antibody) positivity rate of JMT-601 in Part 1 | week 24
Nab (Neutralizing antibody) positivity rate of JMT-601 in Part 1 | week 24
Complete remission rate in Part 2 | week 24, 52, 76, 104
  Complete remission is defined as UPCR (based on 24-hour urine collection) ≤ 0.3, and a stable eGFR (remaining unchanged or decreasing by ≤ 15% compared with the baseline).
Overall remission rate in Part 2 | week 24, 52, 76, 104
  Participants with overall remission are those achieving either complete remission or partial remission. Partial remission is defined as a reduction of proteinuria to 0.3-3.5 g/24 h and 50% lower than baseline with stable renal function.
Relapse rate in Part 2 | week 52, 76, 104
  A relapse is defined as reappearance of UPCR (based on 24-hour urine collection) > 3.5 after complete or partial remission
Time to first complete remission in Part 2 | week 104
Time to first overall remission in Part 2 | week 104
Time to first relapse in Part 2 | week 104
Change of urine protein from baseline in Part 2 | week 12, 24, 52, 76, 104
Change of estimated Glomerular Filtration Rate (eGFR) from baseline in Part 2 | week 12, 24, 52, 76, 104
Immunological response in the anti-PLA2R antibody positive population in Part 2 | week 12, 24, 52, 76, 104
Blood drug concentration of JMT-601 in Part 2 | week 104
ADA (anti-drug antibody) positivity rate of JMT-601 in Part 2 | week 104
Nab (Neutralizing antibody) positivity rate of JMT-601 in Part 2 | week 104
Adverse Events (AEs) in Part 2 | week 104